CLINICAL TRIAL: NCT02510963
Title: An Open-label, Randomized, Controlled Clinical Trial to Determine the Optimal Time for Tenofovir of Anti-HBV Treatment During the Pregnancy Among Chronic HBV-infected Pregnant Women With Normal Liver Function
Brief Title: Optimal Time for Tenofovir Treatment of Anti-Hepatitis B Virus (HBV) During the Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AHCR2014-013
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis B, Chronic
Keywords: Vertical infection transmission; Tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

ARMS (3):
- Tenofovir 24 week (Experimental): Pregnant women with high HBV DNA load in serum and normal liver function were treated with Tenofovir Disoproxil Fumarate 300 mg/day from 24 weeks of gestation to 1 month postpartum
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Tenofovir 28 week (Experimental): Pregnant women with high HBV DNA load in serum and normal liver function were treated with Tenofovir Disoproxil Fumarate 300 mg/day from 28 weeks of gestation to 1 month postpartum
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Tenofovir 32 week (Active Comparator): Pregnant women with high HBV DNA load in serum and normal liver function were treated with Tenofovir Disoproxil Fumarate 300 mg/day from 32 weeks of gestation to 1 month postpartum
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Use Tenofovir at 24week of gestation
  Other Names: Tenofovir
  Arms: Tenofovir 24 week
Drug: Tenofovir Disoproxil Fumarate — Use Tenofovir at 28week of gestation
  Other Names: Tenofovir
  Arms: Tenofovir 28 week
Drug: Tenofovir Disoproxil Fumarate — Use Tenofovir at 32week of gestation
  Other Names: Tenofovir
  Arms: Tenofovir 32 week

SUMMARY:
To determine the optimal time for the Tenofovir treatment of anti-Hepatitis B Virus (HBV) during the pregnancy among women with chronic HBV infection and high HBV DNA load. This is a randomized, open-label, three-arms, parallel-controlled clinical trial. Pregnant women with high HBV load and normal liver function will be treated with tenofovir during the middle or late stage of pregnancy, started from 24th gestational week, 28th gestational week and 32th gestational week through 1 month postpartum, respectively. The HBV DNA load at 40th gestational week of mothers, the intrauterine HBV infection rate of infants will be compared across the three groups.

DETAILED DESCRIPTION:
Tenofovir Disoproxil Fumarate is a American Food and Drug Administration (FDA) pregnancy class B drug. To determine the optimal time for the tenofovir treatment during the pregnancy among women with chronic HBV infection and high HBV DNA load. Pregnant women with high HBV DNA load and normal liver function at second trimester will be randomized into three treatment groups at the 20th week of gestation and treated with tenofovir from 24 weeks, 28 weeks and 32 weeks to 1 month postpartum, respectively. The blood will be drawn at 24 weeks, 28 weeks, 32 weeks, 36 weeks and the delivery, respectively and the HBV DNA load and liver functions will be tested. The status of HBV infection for infants will be observed at 1st month, 7th month and 12th month after the babies were delivered. The HBV DNA load at 40th gestational week of mothers, the intrauterine HBV infection rate of infants and safety outcomes will be compared across the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 40 years old
* Have had HBsAg positive in serum greater than 6 months
* HBV DNA load>10**6 IU/ml
* Gestation week<24 weeks
* Normal liver function
* Able to comprehend and willing to sign the informed consent form

Exclusion Criteria:

* Combined with following infections: hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV), hepatitis E virus (HEV) and human immunodeficiency virus (HIV)
* Got antiviral treatments before 24 weeks of Gestation
* Got immunosuppressor treatment and/or steroids
* Got diagnosis of cirrhosis,hepatocellular carcinoma or severe hepatitis B
* Got serious obstetric complications
* Got evidence of fetal deformity diagnosed by four-dimensional color Doppler ultrasound examination
* Biological father of infant had HBV infection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
HBV DNA load in serum | 40 weeks, from randomization to delivery
  the difference in the percentage of mothers whose HBV DNA load in serum are less than 10*2 IU/ml at delivery among the groups

SECONDARY OUTCOMES:
Intrauterine HBV infection rate of infants | 12 months, from delivery to one-year birth date
  Intrauterine HBV infection rate of infants at the 12th months after delivery
Change in HBV DNA load | 40 weeks, from randomization to delivery
  Total change in HBV DNA load from the start of treatment to the delivery was compared across the three groups
Change in hepatitis B e antigen (HBeAg) titer | 40 weeks, from randomization to delivery
  Total change in HBeAg titer from the start of treatment to the delivery was compared across the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Tianyan Chen, MD,PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China